CLINICAL TRIAL: NCT06469229
Title: Performance Evaluation of Urine DNA Methylation Testing for the Detection of Urothelial Carcinoma in Patients With Hematuria: a Prospective, Multicenter Cohort Study
Brief Title: Performance Evaluation of Urine DNA Methylation Testing for the Detection of Urothelial Carcinoma in Patients With Hematuria
Status: Not yet recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Collaborators: RenJi Hospital (Other); First Hospital of China Medical University (Other); Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TRACE-UC
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Hematuria; Urothelial Carcinoma; Bladder Cancer; Ureter Cancer; Renal Pelvis Cancer
Keywords: Hematuria; Urothelial Carcinoma; Urine DNA Methylation; Multicenter
MeSH Terms: conditions — Hematuria; Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Ureteral Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine sediment DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Urothelial carcinoma (UC) is the most common malignancy of the urinary system. Hematuria is a significant clinical manifestation of UC, often diagnosed through invasive procedures. Urine DNA methylation testing is a promising non-invasive method for early UC detection.

Objectives To evaluate the sensitivity and specificity of urine DNA methylation testing for detecting UC in patients with hematuria, using standard clinical and pathological diagnoses as the gold standard. This study also aim to investigate the association between preoperative urine DNA methylation status and prognosis in UC patients.

For non-UC patients: Follow up for one year to assess the risk of UC development based on preoperative urine DNA methylation status.

Sample Size Calculation Expected sensitivity: 86% Expected specificity: 90% Significance level (Alpha): 0.05 Total participants needed: 1053 (adjusted for 5% dropout rate, 1109 participants will be recruited).

Study Procedure Enrollment and Sample Collection: Screen patients, obtain consent, collect urine samples.

Blinding and Testing: Blinded sample processing and DNA methylation testing. Unblinding and Analysis: Statistical analysis of sensitivity and specificity. Reporting: Compilation and consolidation of clinical trial reports.

Urine DNA methylation testing is expected to demonstrate high sensitivity and specificity for diagnosing urothelial carcinoma (UC) in patients with hematuria. This non-invasive diagnostic method promises to deliver valuable information, potentially leading to improved patient outcomes.

DETAILED DESCRIPTION:
Urothelial carcinoma (UC) is the most common malignancy of the urinary system, and early detection and diagnosis are crucial for patient prognosis. Hematuria is a significant clinical manifestation of UC, but its diagnosis often relies on invasive procedures and imaging, posing a substantial burden on patients. With the advancement of molecular biology techniques, urine DNA methylation testing has emerged as a non-invasive and highly sensitive method for early UC detection. This study aims to evaluate the performance of urine DNA methylation testing in detecting UC in patients with hematuria.

All patients with hematuria will receive standard clinical diagnosis, including examinations, tests, surgeries, and pathological assessments to determine the presence of UC. These clinical diagnoses will serve as the gold standard to evaluate the sensitivity and specificity of urine DNA methylation testing in detecting UC in patients with hematuria.

Based on the expected performance indicators of urine DNA methylation testing and previous study data, the sample size calculation is as follows:

Expected sensitivity: 0.86 Hypothesized sensitivity: 0.80 Expected specificity: 0.90 Hypothesized specificity: 0.85 Significance level (Alpha): 0.05 Considering a dropout rate of 5%, the actual number of participants to be recruited is 1109, ensuring an effective sample size of 1053.

Study Procedure Enrollment and Sample Collection: Screen patients meeting the inclusion criteria, obtain informed consent, collect urine samples, and assign screening numbers. Authorized researchers will perform blinding and aliquoting of the enrolled samples to ensure objectivity and impartiality in the testing process. After blinding, perform urine DNA methylation testing according to the test reagent instructions.

To ensure accuracy and reliability of the results, select a subset of samples with known test results for external methylation sequencing. Authorized researchers will unblind the samples, and the statistical team will analyze the results, calculating sensitivity, specificity, positive predictive value, and negative predictive value of the urine DNA methylation test.

Follow-up:

For UC patients: Evaluate the relationship between preoperative urine DNA methylation levels and postoperative recurrence-free survival, progression-free survival, and overall prognosis.

Clinical Trial Report Each center will compile a clinical summary and submit it to the main center. The main center will consolidate the reports from all centers, draft, and publish the final clinical trial report.

It is anticipated that urine DNA methylation testing will demonstrate high sensitivity and specificity as a non-invasive diagnostic method for detecting urothelial carcinoma (UC) in patients with hematuria. This approach can provide clinicians with crucial reference information, reduce the diagnostic burden on patients, and enhance early detection rates and patient prognosis for UC.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 99 years, with gross or microscopic hematuria (RBC ≥ 3 /HPF or RBC > 18 /μL for men, > 33 /μL for women).
* Able to provide 50ml urine for testing before surgery.
* Consent to participate in the study and sign the informed consent form.

Exclusion Criteria:

* With history of any malignancies (including UC).
* Severe urinary tract infection leading to sepsis.
* Patients with indwelling catheters, nephrostomy, or cystostomy.
* Severe liver or kidney failure or other conditions deemed unsuitable for the study.
* Patients who did not undergo surgical treatment for various reasons.
* Samples with insufficient DNA content or other quality control failures.
* Incomplete clinical or pathological data.
* Patients currently undergoing intravesical or systemic chemotherapy, radiotherapy, immunotherapy, or targeted therapy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective multicenter cohort study aimed at evaluating the effectiveness of DNA methylation biomarkers in detecting urothelial carcinoma in patients with hematuria.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of DNA methylation test in patients with hematuria | 2 weeks
  Evaluate the diagnostic performance of DNA methylation biomarkers by calculating the sensitivity, specificity.

SECONDARY OUTCOMES:
Other diagnostic performance of DNA methylation test in patients with hematuria | 2 weeks
  Calculate the Positive predictive value, negative predictive value，Diagnostic accuracy and the AUROC value of DNA methylation biomarkers.
Comparing the diagnostic performance of of urine DNA methylation and urine cytology | 2 weeks
  Comparing the sensitivity and specificity of urine DNA methylation and urine cytology for the diagnosis of UC in patients with hematuria.
The diagnosis effectiveness of urine DNA methylation test in different types of pathological characteristics of UC | 2 weeks
  Calculate the detection rate of urine DNA methylation test at different tumor grades, invasion depth, tumor size, and tumor number of UC patients
UC patients follow-up | 2 year
  Evaluate the relationship between preoperative urine DNA methylation levels and postoperative progression-free survival in UC patients.
Non-UC patients follow-up | 2 year
  Evaluate the relationship between preoperative urine DNA methylation status and the risk of developing urothelial carcinoma within one year in patients diagnosed as non-UC.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No